CLINICAL TRIAL: NCT00450905
Title: Randomized Evaluation of a Low-Frequency Investigational Device Employing Neuromodulation Therapy in Patients With Fibromyalgia
Brief Title: Pain Relief Investigation of Neuromodulation Therapy in an Adult Fibromyalgia Population
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Fralex Therapeutics (Industry)
Collaborators: PharmaNet (Industry); McDougall Scientific Limited (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F06001
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-02

CONDITIONS: Fibromyalgia; Pain
Keywords: Chronic musculoskeletal pain secondary to Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: PRIMA Device

SUMMARY:
This study is being performed to determine the safety and efficacy of Fralex Neuromodulation Therapy (F-NMT), delivered by the Fralex PRIMA device, in reducing chronic musculoskeletal pain associated with Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic musculoskeletal pain of at least six months duration secondary to FMS using American College of Rheumatology (ACR) criteria and with the minimum of 11 of 18 defined tender points, measured by dolorimeter at a threshold of up to 4 kg of pressure
* Males and females, 18 years and older
* Able to complete assessment index forms unaided by caregiver/interpreter
* Pain score of 4 or greater on the Numerical Rating Scale (NRS), averaged from the Baseline Period scores recorded on the 7 days immediately prior to randomization
* Demonstration of stabilized pain scores as measured on the NRS during the Baseline Period (Days -7 to -1)
* Able to tolerate prohibition of all medications for pain, depression and sleep disorders except for acetaminophen (up to 4 g/day) and cardiac aspirin (up to 325 mg/day) demonstrated for the Stabilization and Baseline Periods prior to randomization
* Able and willing to provide a written informed consent

Exclusion Criteria:

* Unwilling or unable to sign an informed consent, or to comply with the protocol
* Evidence of inflammatory rheumatic disease, secondary fibromyalgia, or other severe painful disorders that might confound assessment of FMS pain
* Currently under treatment (pharmacological or cognitive therapy) for a Major Depressive Episode (MDE) or has demonstrated suicidal ideation in the past
* History or current treatment of migraine, tension or cluster headache requiring regular medication
* History or current treatment of seizure disorder
* History or current treatment of cancer with the exception of basal cell carcinoma and cervical dysplasia
* Cognitive dysfunction or personality disorder which would preclude self-directed treatment, self assessment and / or diary completion
* Clinically significant or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise participation
* Hearing aids, metal implants (excludes dental work) above mid torso or in the cranium (e.g. plates, implants or clips). (Metal implants in parts of the body below mid-torso, such as knee or hips replacements, clips, screws or plates to stabilize fractures are acceptable)
* Pacemakers, defibrillators, implanted neurostimulators, implanted drug pumps or other electrical implanted devices
* Insufficient knowledge of English to complete the self-assessment forms
* History of or current drug or alcohol abuse
* History of abuse of a previous physician relationship or the medical system
* Receiving disability insurance, applying for disability insurance, or engaged in litigation related to FMS
* Use of an investigational drug or device in a controlled study within 30 days
* Pregnancy (U.S. sites only)
* Breastfeeding or intending to breastfeed (U.S. sites only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-03; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Clinically significant pain reduction, evidenced by a statistically significant difference between active and placebo groups in percentage of subjects who achieve a pain reduction of at least 30% at week 12 as compared to the Baseline.

SECONDARY OUTCOMES:
Additional outcome measures will include mood alteration, sleep quality, improvement of physical functioning and relief medication usage by subjects in both groups.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Encinitas, California
  - Garden Grove, California
  - La Jolla, California
  - Lancaster, California
  - Murrieta, California
  - Palmdale, California
  - Gainsville, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Lexington, Kentucky
  - Rochester, Minnesota
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Altoona, Pennsylvania
  - Seattle, Washington
  - Spokane, Washington
- Canada (3):
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario